CLINICAL TRIAL: NCT06178718
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TNP-2092 Capsules, and the Food Effect on the Pharmacokinetics of TNP-2092 Capsules After Single-dose Oral Administration in Healthy Subjects
Brief Title: A Phase 1 Study to Evaluate PK Profile and Food Effects on PK Parameters of TNP-2092 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-2092-01
Record Dates: First submitted 2023-12-07; First posted 2023-12-21 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hyperammonemia
MeSH Terms: conditions — Hyperammonemia | interventions — TNP-2092

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TNP-2092 capsules (Experimental): In single ascending dose study, participants received single oral dose of TNP-2092 capsules 100 to 1200 mg in fasted state.
  In food effect study, participants received single oral dose of TNP-2092 capsules 400 mg in fasted or fed state in a two-sequence, two-period crossover design.
  Interventions: Drug: TNP-2092 capsules
- Placebo (Placebo Comparator): In single ascending dose study, participants received single oral dose of TNP-2092 placebo capsules in fasted state.
  In food effect study, participants received single oral dose of TNP-2092 placebo capsules in fasted or fed state in a two-sequence, two-period crossover design.
  Interventions: Drug: TNP-2092 placebo capsules

INTERVENTIONS:
Drug: TNP-2092 capsules — Administered orally, 100 to 1200 mg
  Other Names: Rifaquizinone
  Arms: TNP-2092 capsules
Drug: TNP-2092 placebo capsules — Administered orally
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The aim of the study was to evaluate the tolerability and pharmacokinetic characteristics of TNP-2092 Capsules after single-dose administration in healthy subjects, and the food effect on pharmacokinetics.

DETAILED DESCRIPTION:
This was a single-center, randomized, double-blind, placebo-controlled, dose-ascending single-dose-administration study, and a study on the food effects on pharmacokinetics. Five dose groups of 100 mg, 200 mg, 400 mg, 800 mg, and 1200 mg will be set up.

The 100 mg, 200 mg, 800 mg, and 1200 mg groups will complete the single ascending dose study, with 10 subjects randomized in each group, 8 subjects receiving TNP-2092 and 2 receiving placebo. The drug will be administered once in each group in the fasting state, and tolerability will be evaluated on D4. Subjects were sequentially enrolled into different dose groups in ascending order of dose, and only when the previous lower dose was confirmed to be safe and well tolerated could they be enrolled into the next higher dose group.

The 400 mg group will complete the single ascending dose study, food effect study and undergo the metabolic transformation evaluation. A total of 18 subjects will be enrolled in the group and randomized into Group A and Group B, with 8 subjects receiving the investigational product and 1 receiving placebo. The drugs will be administered in the fasting state and in the fed state for two cycles, with a wash-out period of 4 days. In terms of the administration sequence, Group A will first take TNP-2092 Capsules or placebo in the fasting state, and then TNP-2092 Capsules or placebo in the fed state; Group B will first take TNP-2092 Capsules or placebo in the fed state, and then TNP-2092 Capsules or placebo in the fasting state. Tolerability evaluation will be conducted on D4 and at the end of the study of food effects on pharmacokinetics (D8).

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female;
* Age: 18-45 years, inclusive;
* BMI: 19.0-26.0 kg/m2, inclusive;
* Female subjects of childbearing potential must agree to practice abstinence or take effective contraceptive measures during the study and at least 70 days (10 weeks) after administration;
* Male subjects must agree to practice abstinence or use condoms as a contraceptive measure during the study and at least 70 days (10 weeks) after administration;
* Subjects whose clinical laboratory test results are within the normal range or whose test results are abnormal, but judged by the investigator to be of no clinical insignificance;
* Those who do not smoke, or have smoked less than 5 cigarettes per day within 3 months before screening; those who do not drink alcohol, or have drunk less than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) within 6 months before screening; those who have not smoked or drunk alcohol within 48 hours before admission to the study site;
* Those who are fully informed of and understand this study, and have signed the Informed Consent Form;
* Those who are willing to follow and able to complete all the study procedures.

Exclusion Criteria:

* Those with symptoms or medical history of cardiovascular, digestive, respiratory, urinary, neurological, blood, immune, endocrine system diseases or tumor, mental illness, or any situation which, in the opinion of the investigator, may threaten the safety of the subjects or affect the correctness of the study results;
* Pregnant or lactating women;
* Those whose blood pressure above 150/90 mmHg or below 85/55 mmHg (supine position);
* Those with regular use of any prescription/over-the-counter drugs, including vitamins, minerals, nutritional supplements or herbs, within 2 weeks before enrollment and during the study;
* Those who are HIV positive, syphilis positive, hepatitis B surface antigen positive, hepatitis C antibody positive, and/or with a positive drug urine test result;
* Those who have a history of alcohol or drug abuse in the past 10 years; Those with an allergic constitution, a history of allergic diseases or a history of drug allergy;
* Those who have had beverages or foods containing methylxanthine (coffee, tea, coke, chocolate and energy drinks), grapefruit (fruit juice) and alcohol within 48 hours (2 days) before the clinical study;
* Those who have taken any drug that changes the activity of liver enzymes within 28 days before taking the investigational product or during the study;
* Those who have donated blood within 3 months before enrollment;
* Those who have participated in any clinical studies within 3 months before enrollment;
* Those who are the staff of the study site directly affiliated to this study or are their immediate family members. Immediate family members are defined as spouses, parents, children or siblings, whether related by blood or legally adopted;
* Those who are employees of TenNor Therapeutics;
* Other circumstances deemed by the investigator to be unsuitable for the subject to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2016-08-02 (Actual); Study Completion 2016-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TNP-2092 Capsules 100mg (Fasting): Participants received single oral dose of TNP-2092 capsules 100mg on Day 1 in fasting state.
- TNP-2092 Capsules 200mg (Fasting): Participants received single oral dose of TNP-2092 capsules 200mg on Day 1 in fasting state.
- TNP-2092 Capsules 400mg - Group A (Fasting - Fed): Participants in TNP-2092 capsules 400mg Group A completed single ascending dose study and food effect study.
  Participants received oral dose of TNP-2092 capsules 400mg on Day 1 in fasting state, and in fed state on Day 5 with a 4-day wash-out period.
- TNP-2092 Capsules 800mg (Fasting): Participants received single oral dose of TNP-2092 capsules 800mg on Day 1 in fasting state.
- TNP-2092 Capsules 1200mg (Fasting): Participants received single oral dose of TNP-2092 capsules 1200mg on Day 1 in fasting state.
- Placebo (Fasting): Participants received TNP-2092 placebo capsules on Day 1 in fasting state, including 2 participants each in 100, 200, 800 and 1200 mg dose group.
- TNP-2092 Capsules 400mg - Group B (Fed -Fasting): Participants received single oral dose of TNP-2092 capsules 400mg on Day 1 in fed state, and in fasting state on Day 5 with a 4-day wash-out period.
- Placebo (Fed-fasting): One participant in 400 mg group B received TNP-2092 placebo capsules on Day 1 in fed state, and in fasting state on Day 5 with a 4-day wash-out period.
- Placebo (Fasting-fed): One participant in 400 mg group A received TNP-2092 placebo capsules on Day 1 in fasting state, and in fed state on Day 5 with a 4-day wash-out period.
Period: Overall Study
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg - Group A (Fasting - Fed) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting) | Placebo (Fasting) | TNP-2092 Capsules 400mg - Group B (Fed -Fasting) | Placebo (Fed-fasting) | Placebo (Fasting-fed)
Started | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 1 | 1
Completed | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TNP-2092 Capsules 400mg - Group A (Fasting-fed): Participants in TNP-2092 capsules 400mg Group A completed single ascending dose study and food effect study.
  Participants received oral dose of TNP-2092 capsules 400mg on Day 1 in fasting state, and in fed state on Day 5 with a 4-day wash-out period.
- Placebo (Fasting): Participants received TNP-2092 placebo capsules on Day 1 in fasting state, including 2 participants each in 100, 200, 800, 1200 mg dose group, and 1 participant in 400 mg group A.
- Placebo (Fed-fasting): Participants received placebo on Day 1 in fed state, and in fasting state on Day 5 with a 4-day wash-out period, including one participant in 400 mg group B.
- Total: Total of all reporting groups
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg - Group A (Fasting-fed) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting) | Placebo (Fasting) | TNP-2092 Capsules 400mg - Group B (Fed -Fasting) | Placebo (Fed-fasting) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 9 | 8 | 1 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 8 | 9 | 8 | 1 | 58
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (9.07) | 33.6 (7.96) | 29.3 (5.34) | 28.9 (10.32) | 25.3 (5.85) | 28.3 (8.72) | 24.9 (5.96) | 19 (0) | 29.1 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 4 | 4 | 3 | 4 | 0 | 24
  Male | 6 | 5 | 4 | 4 | 4 | 6 | 4 | 1 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 8 | 8 | 8 | 9 | 8 | 1 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of TNP-2092 by Assessment of the Number of Participants With Adverse Events (AEs)
Description: To investigate the safety and tolerability of TNP-2092 by assessment of the number of participants with AEs. An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 8 days after the first dosing.
Population: All subjects who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- TNP-2092 Capsules 400mg (Fasting ): Participants received oral dose of TNP-2092 capsules 400mg in fasting state.
- Placebo (Fasting): Participants received TNP-2092 placebo capsules in fasting state.
- TNP-2092 Capsules 400mg - (Fed): Participants received oral dose of TNP-2092 capsules 400mg in fed state.
- Placebo (Fed): Participants received placebo in fed state, with 1 participant in each of the 400 mg groups A and B.
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg (Fasting ) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting) | Placebo (Fasting) | TNP-2092 Capsules 400mg - (Fed) | Placebo (Fed)
Number analyzed (Participants) | 8 | 8 | 16 | 8 | 8 | 10 | 16 | 2
Participants | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 0

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) in Single Ascending Dose Study
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time Frame: Before the first (Day1) administration (within 15 minutes), and 0.5 hour (h), 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h, 16 h, 24 h, 36 h, 48 h and 72 hours (h) after administration
Population: All subjects who have been randomized into groups, have received at least one dose of study drug, and have at least one evaluable pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: h*µg/L
Groups:
- TNP-2092 Capsules 100mg (Fasting); TNP-2092 Capsules 200mg (Fasting); TNP-2092 Capsules 400mg Group A (Fasting); TNP-2092 Capsules 800mg (Fasting); TNP-2092 Capsules 1200mg (Fasting): Participants received single oral dose of TNP-2092 in fasting state.
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg Group A (Fasting) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
h*µg/L | 67.9 (29.9) | 164 (65.7) | 201 (71.4) | 408 (480) | 339 (176)

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 to the Last Measurable Concentration (AUC0-last) in Single Ascending Dose Study
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma PK parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*µg/L
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg Group A (Fasting) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
h*µg/L | 65.4 (28.8) | 161 (65.0) | 197 (71.0) | 404 (478) | 335 (175)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of TNP-2092 in Single Ascending Dose Study
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg Group A (Fasting) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
µg/L | 16.7 (7.80) | 41.7 (17.9) | 48.5 (20.8) | 97.4 (117) | 70.3 (41.2)

5. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of TNP-2092 in Single Ascending Dose Study
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg Group A (Fasting) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
h | 3.76 (0.46) | 3.50 (0.53) | 3.50 (1.20) | 3.75 (1.04) | 3.25 (1.17)

6. Primary Outcome: Terminal Elimination Half-life (T1/2) in Single Ascending Dose Study
Description: as for outcome 3
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg Group A (Fasting) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
h | 2.348 (1.0494) | 2.778 (1.1949) | 2.553 (1.2619) | 2.819 (0.8444) | 3.278 (1.1161)

7. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) in Food Effect Study
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*µg/L
Groups:
- TNP-2092 Capsules 400mg (Fasting): Participants in TNP-2092 capsules 400mg Group A and Group B received single oral dose of TNP-2092 capsules 400 mg in fasting state.
- TNP-2092 Capsules 400mg (Fed): Participants in TNP-2092 capsules 400mg Group A and Group B received single oral dose of TNP-2092 in fed state.
Arm/Group | TNP-2092 Capsules 400mg (Fasting) | TNP-2092 Capsules 400mg (Fed)
Number analyzed (Participants) | 16 | 16
h*µg/L | 214 (91.7) | 632 (349)

8. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From 0 to the Last Measurable Concentration (AUC0-last) in Food Effect Study
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*µg/L
Groups:
- TNP-2092 Capsules 400mg (Fasting): Participants in TNP-2092 capsules 400mg Group A and Group B received single oral dose of TNP-2092 in fasting state.
Arm/Group | TNP-2092 Capsules 400mg (Fasting) | TNP-2092 Capsules 400mg (Fed)
Number analyzed (Participants) | 16 | 16
h*µg/L | 211 (90.6) | 628 (349)

9. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of TNP-2092 in Food Effect Study
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | TNP-2092 Capsules 400mg (Fasting) | TNP-2092 Capsules 400mg (Fed)
Number analyzed (Participants) | 16 | 16
µg/L | 50.2 (25.2) | 102 (36.6)

10. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of TNP-2092 in Food Effect Study
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 400mg (Fasting) | TNP-2092 Capsules 400mg (Fed)
Number analyzed (Participants) | 16 | 16
h | 3.56 (0.89) | 6.94 (2.72)

11. Primary Outcome: Terminal Elimination Half-life (T1/2) in Food Effect Study
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 400mg (Fasting) | TNP-2092 Capsules 400mg (Fed)
Number analyzed (Participants) | 16 | 16
h | 2.74 (1.24) | 3.69 (0.98)

ADVERSE EVENTS:
Time Frame: Up to 8 days after the first dosing.
Arm/Group | TNP-2092 Capsules 100mg (Fasting) | TNP-2092 Capsules 200mg (Fasting) | TNP-2092 Capsules 400mg (Fasting ) | TNP-2092 Capsules 800mg (Fasting) | TNP-2092 Capsules 1200mg (Fasting) | Placebo (Fasting) | TNP-2092 Capsules 400mg - (Fed) | Placebo (Fed)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/16 | 0/8 | 0/8 | 0/10 | 0/16 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/16 | 0/8 | 0/8 | 0/10 | 0/16 | 0/2
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 2/16 | 1/8 | 1/8 | 1/10 | 2/16 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNP-2092 Capsules 100mg (Fasting) (N=8) | TNP-2092 Capsules 200mg (Fasting) (N=8) | TNP-2092 Capsules 400mg (Fasting ) (N=16) | TNP-2092 Capsules 800mg (Fasting) (N=8) | TNP-2092 Capsules 1200mg (Fasting) (N=8) | Placebo (Fasting) (N=10) | TNP-2092 Capsules 400mg - (Fed) (N=16) | Placebo (Fed) (N=2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT06178718/Prot_SAP_000.pdf